CLINICAL TRIAL: NCT06272357
Title: Clinical Audit on the Use of Antiarrhythmic Drugs in Pediatric Age Group
Brief Title: The Use of Antiarrhythmic Drugs in Pediatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Abdel-Aziz mohamed, Principal Investigator, Assiut University
Other Study IDs: Antiarrhythmic drugs
Record Dates: First submitted 2023-11-23; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Antiarrhythmic Drug Adverse Reaction
MeSH Terms: interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antiarrhythmic drugs — Antiarrhythmic drugs in pediatrics

SUMMARY:
A study on the use of antiarrhythmic drugs in pediatric age group, in Assiut University Children's Hospital, a clinical audit

DETAILED DESCRIPTION:
Arrhythmias occur in children and adolescents with congenital heart disease as well as those with structurally normal hearts.

Rhythm disturbances (arrhythmias) are not uncommon in sick children admitted in pediatric intensive care unit. These occur as a result of abnormalities in, or insults to, the cardiac conduction system or heart tissues. A rhythm disturbance in a child should be treated as life threatening emergency.

The generation of the action potential and the regional differences that are observed throughout the heart are the result of the selective permeability of ion channels distributed on the cell membrane.

Abnormalities in surface membrane ion channel function are central to arrhythmogenesis.

Antiarrhythmic medications primarily affect the ion channels in cardiac myocytes that are responsible for generating currents that create the action potential.

By altering the activity of these ion channels, the action potential is changed to reduce the likelihood of sustained arrhythmias.

These drugs are predominantly used in treatment of arrhythmia but in addition they are also used as a treatment of other cardiac and non-cardiac conditions.

For example, Calcium channel blockers have been one of the most widely used classes of antihypertensive agents in the last 20 years.

Carvedilol (a beta blocker agent) can be safely used for treatment of chronic heart dysfunction in pediatric patients with dilated cardiomyopathy.

β-blockers are also an essential component of pharmacologic therapy for children with congestive heart failure.

There is a wide range of antiarrhythmic drugs used in treatment of arrhythmias. The modernized comprehensive classification of both established and potential antiarrhythmic drugs was proposed in 2018 Class 0: HCN channel-mediated pacemaker current (If) block Class I: Antiarrhythmic that affect sodium channels (slow depolarization) Class II: Drugs that counteract the sympathetic nervous system, predominantly beta-blockers Class III: drugs that affect the potassium channels (prolong repolarization) Class IV: Drugs that affect calcium channels (Calcium channel blockers) Class V: mechanically sensitive ion channels, Mechanosensitive channel blockers Class VI: Gap junction channel blockers Class VII: Upstream target modulators.

In this study the aim is to describe the use of Cardiovascular Drugs in Pediatric Cardiology unit Assiut University. As regard: indications of use, proper dosage and proper management of side effects of their use.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with Arrhythmic cardiac diseases admitted at cardiology unit Assiut University Hospital aged from 1 month to 18 years.
* All patient receiving antiarrhythmic drugs admitted to Assiut University Hospital for Children.

Exclusion Criteria:

• Any patient on drugs other than antiarrhythmics.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Patients with Arrhythmic cardiac diseases admitted at cardiology unit Assiut University Hospital aged from 1 month to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Detect the rate of use of antiarrhythmic drugs in pediatrics and the different indications for them other than the control of arrhythmia. | Baseline
  A study on the use of antiarrhythmic drugs in pediatric age group, in Assiut University Children's Hospital and the different indications for them other than the control of arrhythmia